CLINICAL TRIAL: NCT04915547
Title: Efficacy of Group Exercise Program on Pain and Disability in Older People With Nonspecific Low Back Pain: Feasibility of a Randomized Controlled Trial.
Brief Title: Efficacy of Group Exercise Program in Older People With Nonspecific Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of the Valleys of Jequitinhonha and Mucuri (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 30042021
Record Dates: First submitted 2021-05-15; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: Low Back Pain; Back Pain
MeSH Terms: conditions — Low Back Pain; Back Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-Based Exercise (Experimental): The group-based exercise (GBE) programme will be delivered by a physiotherapist. The GBE comprises three sessions per week of group-based exercise in a local community centre, for 8 weeks.
  Interventions: Other: Group-Based Exercise
- Control Group (No Intervention): Participants randomly allocated to the control group will remain on a waiting list. In addition, weekly contact will be made to ensure that they do not start treatment during the study protocol. After the end of the study, participants randomly allocated to the control group will receive the same intervention as the Group-Based Exercise.

INTERVENTIONS:
Other: Group-Based Exercise — Each group session will consist of 10 to 18 participants and each exercise session will last 60 minutes and consist of four stages: (1) five minutes warm up (i.e. self-regulated walk); (2) twenty minutes of moderate intensity walking (3) thirty minutes of resistance training for the major muscles of the leg, trunk and arm and balance exercises that progress in difficulty; (4) five-minute cool down period (i.e. self-regulated walk). The exercise intensity will be assessed by one of the following criteria: 1) Resistance training - Point of volitional fatigue. Walking - Somewhat difficult (Borg at 3 to 4). The intensity will be increased according to the ACSM guideline.
  The exercise was set up based on changes in instruments of evaluation of the older peoples as, Berg Balance Scale; Dynamic Gait Index and Timed Up and Go. In addition, exercises commonly used in primary health care groups. The protocol will take place in a gymnasium and will be supervised by a trained instructor.
  Arms: Group-Based Exercise

SUMMARY:
The main objective of the study is to assess the feasibility of a randomized clinical trial that investigates the effects of an 8-week group exercise program on pain, disability, fear of falling, overall impression of recovery, frequency of falls and level of physical activity in elderly people with nonspecific low back pain.

DETAILED DESCRIPTION:
The main objective of the study is to assess the feasibility of a randomized clinical trial that investigates the effects of an 8-week group exercise program on pain, disability, fear of falling, overall impression of recovery, frequency of falls and level of physical activity in elderly people with nonspecific low back pain. The evaluation of feasibility will be related to: (1) blinding the evaluator to allocate the groups; (2) eligibility and recruitment rates; (3) acceptability of random allocation to a group; (4) possible contamination between groups; (5) adherence to treatment; (6) satisfaction with the treatment; and (7) difficulty in understanding the information provided by the physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* Older people aged 60 years old or over who have nonspecific LBP, defined as pain below the costal margin and above the lower gluteal folds, with or without referred leg pain for at least 3 months.
* Disability with score 4/24 in Roland-Morris Disability Questionnaire or higher and persistent back pain of pain 3/10 or higher.

Exclusion Criteria:

* Suspected or confirmed serious spinal pathology (fracture, metastatic, inflammatory or infective diseases of the spine, cauda equina syndrome/widespread neurological disorder);
* Radiculopathy (i.e. presence of 2 of the 3 following criteria: strength, reflex or sensation alterations compatible with lumbosacral nerve root compression);
* Previous history of spinal surgery; scheduled for major surgery during the study or at the follow up period;
* Any of the contraindications to exercise listed on page 103 of the American College of Sports Medicine (ACSM) guidelines.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of blinding the assessor | 8 weeks from randomization
  Feasibility of blinding will be assessed by asking the assessor two questions at the end of the follow-up assessment:
  1. Did you receive any information that indicated to you which group the participant was assigned to?
  2. How did you receive information about group assignment?
  Assessor's guess regarding group assignment group will be recorded for each participant.
  The responses will be coded as correct or incorrect guess.
  The frequency and relative rates of 'Yes' and 'No' as the answer to the first question will be computed, as will the frequency and relative rates of correct and incorrect guesses. Finally, reasons for guesses will be recorded as verbatim and reported.
Eligibility and recruitment rates | 8 weeks from randomization
  Eligibility and recruitment rates
Acceptability of random allocation to a treatment group | 8 weeks from randomization
  Outcome assessor will ask the participants if random allocation to one of the two treatment groups is acceptable to the participants. Responses will be recorded as 'Acceptable', 'Not acceptable' or 'No preference'.
  The frequencies of each response will be computed separately for each treatment condition.
Understanding possible contamination between the groups | 8 weeks from randomization
  Measures to assess:
  Have you talked to other participants in this study about the intervention they are receiving? Has your attitude towards the intervention changed after talking to the participant (s) in the other group? Are any of the participants in the other group aware of the type of intervention you are receiving in this study?
  The frequencies of the participants who responded affirmatively to each question will be computed separately for each treatment condition.
Adherence to treatment | 8 weeks from randomization
  Adherence to treatment measured by frequency during the intervention
Satisfaction with the treatment | 8 weeks from randomization
  All the participants of the intervention group will be asked to respond an adapted version of the MedRisk Instrument for Measuring Patient Satisfaction With Physical Therapy Care at 1 week following treatment. The question asked will be:
  1. Did my physiotherapist carefully explain the treatments I received?
  2. Did my physiotherapist treat me respectfully?
  3. Did my physiotherapist answer all my questions? n general, am I completely satisfied with the services I received from my physical therapist? Responses to this question are made on a five-point categorical scale 1='completely disagree'; 2='Disagree'; 3= 'Neutral'; 4=' Agree'; 5=' Completely agree').
  The frequency of response for each question will be analyzed
Difficulty in understanding the information provided by the physiotherapist | 8 weeks from randomization
  Difficulty in understanding the information provided by the physiotherapist measured on a five-point categorical scale: Very easy, Easy, Neither easy nor difficult, Difficult, Very difficult

SECONDARY OUTCOMES:
Pain intensity | 8 weeks from randomization
  Pain intensity measured with a Numerical Rating Scale from 0 to 10, , where 0 does not cause pain and 10 is the worst pain imaginable.
Disability | 8 weeks from randomization
  Disability measured with the Roland-Morris Disability Questionnaire. The questionnaire has 24 items with scores of 0 or 1 (yes or no) and the total ranges from zero (suggesting no disability) to 24 (severe disability).
Fear of falling | 8 weeks from randomization
  Fear of falling measured with the Falls Efficacy Scale- International. The Falls Efficacy Scale - International presents questions about the concern with the possibility of falling when performing 16 activities, with respective scores from one to four. The total score can range from 16 (no concern) to 64 (extreme concern).
Level of physical activity | 8 weeks from randomization
  Level of physical activity measured with the Physical Activity Rating scale. It is a progressive scale with scores from 0 to 7, in which the most appropriate option for the history of physical activity practice in the last 30 days should be selected.
Global perception of recovery | 8 weeks from randomization
  Global perception of recovery measured with Global Effect Perception Scale. This is a numerical scale where -3 represents "worse than ever", 0 "without modification" and 3 "completely recovered". A higher score means greater recovery from the condition.
Frequency of falls | 8 weeks from randomization
  Frequency of falls assessed by the number of falls during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Letícia Soares Fonseca, Principal Investigator — Federal University of the Valleys of Jequitinhonha and Mucur

IPD SHARING:
Plan to Share IPD: No